CLINICAL TRIAL: NCT00006224
Title: Evaluation of Gemcitabine in Persistent or Recurrent Non-Squamous Cell Carcinoma of the Cervix
Brief Title: Gemcitabine in Treating Patients With Persistent or Recurrent Cancer of the Cervix
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000068144; GOG-0128F
Record Dates: First submitted 2000-09-11; First posted 2003-11-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2005-06

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Gemcitabine

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine in treating patients who have persistent or recurrent cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of gemcitabine in patients with persistent or recurrent nonsquamous cell carcinoma of the cervix who failed higher priority treatment protocols.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes weekly for 3 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: Approximately 15-37 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of persistent or recurrent nonsquamous cell carcinoma of the cervix that has failed local therapeutic measures and is considered incurable

  * Eligible subtypes:

    * Adenocarcinoma
    * Adenosquamous carcinoma
    * Undifferentiated carcinoma
  * Must have documented disease progression
  * Histologic confirmation of original primary tumor required
* Bidimensionally measurable disease
* Ineligible for higher priority GOG protocol

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 100,000/mm^3
* Granulocyte count at least 1,500/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT and alkaline phosphatase no greater than 3 times normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* No significant infection
* Not pregnant
* Fertile patients must use effective contraception
* No other invasive malignancy within the past 5 years except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent filgrastim (G-CSF)

Chemotherapy:

* No prior gemcitabine
* At least 3 weeks since other prior chemotherapy for cervical cancer and recovered
* No more than 1 prior chemotherapy regimen (single or combination cytotoxic therapy)

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy for cervical cancer and recovered

Surgery:

* At least 3 weeks since prior surgery for cervical cancer and recovered

Other:

* No prior cancer treatment that would preclude study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Primary Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell J. Schilder, MD, Study Chair — Fox Chase Cancer Center
Locations (39):
- United States (38):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Tufts University School of Medicine, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Schilder RJ, Blessing J, Cohn DE. Evaluation of gemcitabine in previously treated patients with non-squamous cell carcinoma of the cervix: a phase II study of the Gynecologic Oncology Group. Gynecol Oncol. 2005 Jan;96(1):103-7. doi: 10.1016/j.ygyno.2004.09.027. PMID 15589587